CLINICAL TRIAL: NCT04890002
Title: Improving Sleep With the Far-infrared Emitting Pyjamas: A Pilot Randomized Controlled Trial
Brief Title: Improving Sleep With the Far-infrared Emitting Pyjamas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Dr, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFEP
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Far-infrared emitting pyjamas (FIR pyjamas) group (Experimental): Subjects in this group will be provided the Far-infrared emitting pyjamas. The FIR pyjamas was fabricated by using two textile materials, pure cotton fibres and the proposed man-made FIR fibres with the far-infrared emitting function.
  Interventions: Device: Far-infrared emitting pyjamas
- Sham-pyjamas Group (Sham Comparator): To control the placebo effect in the FIR pyjamas group, participants in this group will receive pyjamas with identical physical appearance which are produced using the same fabrication process as the pyjamas received in FIR pyjamas group. The sham-pyjamas are made of pure cotton fibres and man-made fibres without the far-infrared emitting function. The participants will be asked to wear the sham-pyjamas daily at night for 6 consecutive weeks.
  Interventions: Device: Sham-pyjamas

INTERVENTIONS:
Device: Far-infrared emitting pyjamas — Clothing made in far infrared (FIR) - based textiles could be a sustainable way for alleviating sleep problems with many advantages. Firstly, the proposed far infrared textiles are made of man-made profiled fibers without the addition of chemicals such as ceramic additives or other related coatings.
  Arms: Far-infrared emitting pyjamas (FIR pyjamas) group
Device: Sham-pyjamas — The sham-pyjamas are made of pure cotton fibres and man-made fibres without the far-infrared emitting function.
  Arms: Sham-pyjamas Group

SUMMARY:
The aim of this study is to explore the effects of a far-infrared emitting pyjamas on improving sleep in adults with poor sleep.

DETAILED DESCRIPTION:
Objectives: To explore the effects of a far-infrared emitting pyjamas on improving sleep in adults with poor sleep.

Hypothesis: Subjects who wear the far-infrared emitting pyjamas (FIR pyjamas) will have greater improvement in sleep quality than the subjects in sham pyjamas control group (sham-pyjamas) at 2, 4 and 6 weeks.

Design and subjects: A pilot randomized sham-controlled trial. Subjects with subjective sleep complaints will be recruited from the community. 40 subjects will be randomized to far-infrared emitting pyjamas and sham-pyjamas groups in a 1: 1 ratio. Study instrument: Pittsburgh Sleep Quality Index (PSQI) will be used as an overall evaluation of sleep quality.

Interventions: Subjects in the FIR pyjamas group will received pyjamas with far-infrared emitting features and will wear it every night for 6 weeks; subjects in the sham-pyjamas group will receive pyjamas in identical appearance without far-infrared emitting features.

Outcome measures: The primary outcome measure is the PSQI score. Other measures include insomnia severity index (ISI), sleep parameters derived from 7-day sleep diary, Hospital Anxiety and Depression Scale (HADS), Epworth Sleepiness Scale (ESS) and Satisfaction With Life Scale (SWLS) at 2, 4 and 6 weeks. Acceptability of the far-infrared emitting pyjamas will also be evaluated.

Data Analysis: Differences in the questionnaire scores, subjective sleep parameters will be examined using a mixed-effects model. Clinical significance of sleep improvement between two groups will be compared with chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Hong Kong residents who are able to read Chinese;
* Aged 18 - 65 years;
* Subjective sleep complaints of having difficulties in falling asleep, difficulties in staying asleep, or early morning awakening with consequences for daily life for at least 3 months.
* Pittsburgh Sleep Quality Index total score of at least 5 indicating sleep disturbance with 89.6% sensitivity and 86.5% specificity; and
* Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

* Currently receiving psychotherapy or participating in other clinical trials for insomnia;
* Pregnancy;
* Shift workers;
* At significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (score ≥ 3);
* No comorbid sleep disorders primarily requiring other treatment, such as sleep apnea or narcolepsy; and
* Taking herbal remedies, over-the-counter medication, or psychotropic drugs that target insomnia within the 2 weeks prior to baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 2, week 4, and week 6
  The PSQI is a self-reported evaluation of the overall sleep quality. Subjects will be asked to report the sleep parameters of their sleep problem, use of sleep medicine, disturbance, and daytime dysfunction with 0-3 rating. The time frame of PSQI adopted in this study will be changed from "past 1 month" to "past 2 weeks". The PSQI is a reliable and validated tool widely used in sleep studies.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, week 2, week 4, and week 6
  The ISI is a seven-item self-rating scale. The subjects rate the severity of insomnia, the distress, and the functional impairment associated with insomnia on a 5-point Likert scale. The ISI is a validated instrument which has been commonly used in clinical trials of insomnia.
The 7-day daily sleep diary | Baseline and week 6
  The standardized sleep diary records the bedtime and rising time, from which the total time in bed (TIB) can be calculated. Subjects will be asked to estimate sleep-onset latency, wake after sleep onset, and total sleep time (TST). They will also rate their sleep quality on a 4-point scale (very good, fairly good, fairly bad, and very bad).
Hospital Anxiety and Depression Scale (HADS) | Baseline, week 2, week 4, and week 6
  The HADS is a 14-item self-administrated questionnaire, which assess the severity of depressive and anxiety symptoms
Epworth Sleepiness Scale (ESS) | Baseline, week 2, week 4, and week 6
  The ESS is a self-rated questionnaire assessing the level of daytime sleepiness in eight common daily activities. The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. The questionnaire takes no more than 2 or 3 minutes to answer.
The 5-item Satisfaction with Life Scale (SWLS) | Baseline, week 2, week 4, and week 6
  The score of SWLS is found to predict mental health which has been used for assessing subjective well-being of subjects with health conditions. Scores consist of a raw score (between 5 and 35). Higher scores represent higher life satisfaction. Scorers can be assigned into six well-being categories and interpretative text in provided for each.
Multidimensional Fatigue Inventory (MFI) | Baseline, week 2, week 4, and week 6
  MFI is a 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. In an initial psychometric evaluation, developers reported an internal consistency ranging from .53 to .93. The scale was also found to be sensitive to differences between the participant groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wing Fai YEUNG, Dortor, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Wing Fai YEUNG, Hong Kong, Hong Kong